CLINICAL TRIAL: NCT07276932
Title: Clinical Study on Acupoint Application Based on the Theory of "State-target Syndrome Differentiation" in Relieving qi Deficiency and Constipation in Patients With Colorectal Cancer Undergoing Postoperative Chemotherapy
Brief Title: Clinical Study of Acupoint Application on Relieving qi Deficiency and Constipation in Patients Undergoing Chemotherapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2025-0322
Record Dates: First submitted 2025-11-17; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-01

CONDITIONS: Postoperative Chemotherapy; Chemotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupoint application + conventional treatment and nursing program (Experimental)
  Interventions: Drug: Acupoint application; Behavioral: Routine treatment and nursing of constipation
- Routine treatment and nursing of constipation (Active Comparator)
  Interventions: Behavioral: Routine treatment and nursing of constipation

INTERVENTIONS:
Drug: Acupoint application — 1. The traditional Chinese medicine patch was prepared according to the ratio of astragalus: tangerine peel: sesame seed seed: white mustard seed = 6:6:2:1, and an appropriate amount of honey was used to make the shape.
  2. Timing of application: finger time (6:30 am).
  3. Acupoint prescription: Zusanli (bilateral), Zhongwan (CV 12), Qihai (CV 6) and Guanyuan (CV 4).
  4. Location of acupoint: the patient went to the supine position or sitting position with knee flexion. Zusanli (Zusanli) is three cun below the outer knee of both lower limbs; Zhongwan (CV 12) is located from xiphoid process to navel midpoint. Qihai acupoint is located on the median line of the human abdomen, three transverse fingers down from the umbilicus. Location of Guanyuan point: 3 cun (four fingers) below the belly button.
  5. Treatment time and frequency: once a day, 2 hour
  Arms: Acupoint application + conventional treatment and nursing program
Behavioral: Routine treatment and nursing of constipation — 1. Diet care: supplement adequate dietary fiber and adequate water intake.
  2. Defecation training: regular defecation training in the morning. Patients or their family members should massage the abdomen clockwise for more than 10 minutes every day to increase the amount of activity.
  3. Emotional nursing: explain disease-related knowledge, improve patients' understanding of constipation, relieve bad emotions in time, help patients build confidence and actively participate in treatment.

SUMMARY:
4.1 Research Content

1. Clarifying the acupoint application scheme for deficiency and constipation in CRC patients undergoing chemotherapy: the preliminary acupoint application scheme for deficiency and constipation in CRC patients was formulated according to the systematic literature search, analysis of acupoint and traditional Chinese medicine prescription, analysis of meridian tropism of acupoints, Chinese herbal medicine taste and meridian tropism, etc., and multidisciplinary expert consultation. Through two rounds of Delphi expert letter consultation, the acupoint application scheme for deficiency and secret of CRC patients undergoing chemotherapy was determined.
2. Randomized controlled trials were conducted to compare the effect of acupoint application scheme and conventional treatment in improving constipation symptoms, total clinical efficacy, and improving patient comfort rate in CRC patients undergoing chemotherapy.

4.2 Key problems to be solved Based on the theory of "state-target dialectics", the analysis of acupoints and traditional Chinese medicine prescriptions, the analysis of meridian tropism of acupoints, the flavor and meridian tropism of Chinese herbs are used to select Chinese herbs that moisten the intestine and relieve defecation, strengthen the central and qi, and explore the acupoint application to provide a basis for more effective application of acupoint application in the treatment of qi deficiency and constipation in patients with CRC chemotherapy, form a generalized integrated Chinese and western medicine diagnosis and treatment plan, and promote the development of integrated Chinese and western medicine.

4.3 Expected Goals

1. Clarify the diagnosis and treatment plan of acupoint application in the treatment of qi deficiency and constipation in patients with colorectal cancer.
2. The flexible application of classic formula and scientific acupoint selection and sticking can effectively relieve qi deficiency and constipation in CRC patients undergoing chemotherapy, improve the total clinical efficacy and comfort of patients. It has been used in clinical practice and promoted to other medical institutions.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of colorectal cancer
2. Chemotherapy was performed after surgery
3. Diagnosis of qi deficiency and constipation
4. Age ≥18 years old

Exclusion Criteria:

1. Clinical diagnosis of other digestive tract or anal organic diseases
2. Observed with severe cardiac, hepatic, renal insufficiency or other complications
3. Allergic constitution or allergy to a drug in constipation paste

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2025-07-16 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The Nimodipine method was used to calculate the total symptom score of patients | Five days after the intervention
  Efficacy index =[(pre-treatment score - post-treatment score)/pre-treatment score]× 100%, which was divided into 4 grades: clinical cure, marked effect, effective and ineffective. Clinical recovery: the main symptoms and signs disappeared or basically disappeared, and the efficacy index was ≥ 95%. Marked efficacy: the main symptoms and signs were significantly improved, 70% ≤ efficacy index < 95%; Effective: the main symptoms and signs were significantly improved, 30% ≤ efficacy index < 70%; Ineffective: the main symptoms and signs were not significantly improved, or even aggravated, and the efficacy index was less than 30%.
Constipation symptom assessment form | Before and after 5 days of intervention
  It was formulated by the Anorectal Surgery Group of Chinese Society of Surgery of Chinese Medical Association, and included six dimensions: defecation frequency, defecation time, defecation difficulty, stool character, abdominal distension, falling, incomplete and fullness. A 4-point scale was used to evaluate the severity of symptoms.The higher the score, the more severe the constipation symptoms.The minimum score was 0 and the maximum score was 18.

SECONDARY OUTCOMES:
Chinese version of Symptom Checklist for Constipation (PAC-SYM) | Before and after 5 days of intervention
  Developed by MaPi Research Trust in France, it has good reliability and validity and has been widely used in clinical practice. The questionnaire included 3 dimensions and 12 items, including stool shape, rectal and abdominal symptoms, etc. The severity of symptoms was evaluated using a 5-point scale. The higher the score, the more severe the patient's constipation symptoms. The lowest score was 0 and the highest score was 48.
Constipation quality of life self-rating scale (PAC-QOL) | Before the intervention and 5 days after the intervention
  The Chinese version was developed by Mapi Research Trust, with 28 items in total, involving patients' physiology, social psychology, worry, satisfaction and other aspects (see Appendix 3). It can comprehensively measure the quality of life of patients with constipation, and objectively and truly reflect the patient's status, treatment satisfaction and acceptance. A higher score indicates a higher level of quality of life in patients with constipation. The lowest score was 28 and the highest score was 112.
TCM syndrome rating scale of qi deficiency and constipation | Before the intervention and 5 days after the intervention
  The application was developed by Li Jinyue et al., which reflected the symptoms of TCM syndromes, including shortness of breath, defecation weakness, lack of breath and lazy speech, and sweating. According to the patient's description of the related symptoms, the degree of severity was evaluated and divided into four levels: none, mild, moderate, and severe, and scored 0, 1, 2, and 3 points respectively. The higher the score, the more severe the patient's qi deficiency and constipation symptoms. The lowest score was 0 and the highest score was 12.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China